CLINICAL TRIAL: NCT02364453
Title: The Effect of Histamine H1 Receptor Antagonist, Clemastin, on PACAP38 Induced Headache in Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Song Guo (Other)
Responsible Party: Sponsor-Investigator, Song Guo, Medical Doctor, PhD.-student, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H-4-2014-103
Record Dates: First submitted 2014-10-07; First posted 2015-02-18 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo to PACAP38 (Experimental): Pre-treatment with placebo. PACAP38 8pmol/kg/min
  Interventions: Drug: PACAP38
- Clemastin 1 mg/ml to PACAP38 8pmol/kg/min (Experimental): Pre-treatment with Clemastin 1 mg/ml PACAP38 8 pmol/kg/min
  Interventions: Drug: PACAP38

INTERVENTIONS:
Drug: PACAP38 — Giving doses of 4, 6 or 8 pg/kg/min on three separate trial days.
  Other Names: Pituitary Adenylate Cyclase Activating Peptide 38

SUMMARY:
The purpose of this study is to determine the effects of antihistamine (Clemastin) on migraines triggered by pituitary adenylate cyclase activating peptide-38 (PACAP38) as well as on biochemical markers for mast cell degranulation in migraine patients. Also, to investigate the occurrence of migraine in migraine patients after infusion of PACAP38 in lower dosages than previously investigated. As this has never been done before it is unknown how a lower dose of PACAP38 will affect 1) the incidence of migraine attacks, 2) the accompanying symptoms, 3) head pain characteristics, and 4) debut and duration of migraine attacks.

Our three hypotheses are:

1. Pre-treatment with Clemastin reduces PACAP38 sensitivity and inhibits development of migraine in migraine patients.
2. Clemastin inhibits the increase in plasma concentration of TNF-alpha, histamine and tryptase after PACAP38-infusion.
3. PACAP38 in lower dosages (4, 6 and 8 pmol/kg/min) induces migraine in migraine patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of antihistamine (Clemastin) on migraines triggered by pituitary adenylate cyclase activating peptide-38 (PACAP38) as well as on biochemical markers for mast cell degranulation in migraine patients. Also, to investigate the occurrence of migraine in migraine patients after infusion of PACAP38 in lower dosages than previously investigated. As this has never been done before it is unknown how a lower dose of PACAP38 will affect 1) the incidence of migraine attacks, 2) the accompanying symptoms, 3) head pain characteristics, and 4) debut and duration of migraine attacks.

ELIGIBILITY:
Inclusion Criteria:

* migraine patients fulfilling IHS criteria for migraine without aura, ages 18-50, 50-100 kg, fertile women must be using safe prevention

Exclusion Criteria:

* other types of primary headache than migraine
* headache on trial day or later than 48 hours before trial day
* migraine up to three days before trial day
* any type of cardiovascular disease
* clinical signs or patient history of any type of illness that the medical doctor in charge of trials deems relevant for participation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Development of migraine in migraine patients | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Professor, Study Director — Danish Headache Center
Locations (1):
- Danish Headache Center & Department of Neurology, Copenhagen, Glostrup, Denmark